CLINICAL TRIAL: NCT01857245
Title: Intensive Models of HCV Care for Injection Drug Users
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Prisma Health-Upstate (Other)
Collaborators: Clemson University (Other); Albert Einstein College of Medicine (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 1R01DA034086-01, 2011-555; 1R01DA034086-01 (NIH)
Record Dates: First submitted 2013-05-16; First posted 2013-05-20 (Estimated); Results first posted 2025-02-03 (Actual); Last update posted 2025-02-03 (Actual); Status verified 2018-06

CONDITIONS: Hepatitis C; Medication Adherence
Keywords: addiction; Adherence (attribute); Adverse effects; Agonist; Antiviral Agents; arm; base; care delivery; Caring; Chronic Hepatitis C; Clinic; Clinical Trials; Complex; Computer Simulation; cost; cost effective; cost effectiveness; Data; Development; Directly Observed Therapy; Disease; Dose; Drug resistance; drug resistant virus; Educational aspects; Epidemic; experience; Frequencies (time pattern); Fright; Genotype; Group Therapy; Health Care Costs; Health Personnel; Healthcare Systems; Hepatitis C; Hepatitis C Prevalence; Hepatitis C Transmission; Hepatitis C virus; HIV; Homelessness; improved; Incidence; Infection; Injecting drug user; Injection of therapeutic agent; Intensive Care; Interferons; Intervention; Knowledge; Life; Liver diseases; Liver Failure; liver transplantation; Living Costs; Mental disorders; Methadone; methadone clinic/center; Modeling; Mortality Vital Statistics; Motivation; multidisciplinary; Opiates; Oral; Outcome; Patients; Persons; Pharmaceutical Preparations; Physicians; pill (pharmacologic); Play; Poverty; Primary Health Care; programs; Psychiatric therapeutic procedure; psychosocial; Publishing; Quality-Adjusted Life Years; Randomized; Randomized Controlled Trials; randomized trial; Recruitment Activity; Regimen; Resistance; Resistance development; response; Risk; risk perception; Role; Site; skills; Social support; standard care; substance abuse treatment; success; Time; Treatment outcome; Treatment Protocols; treatment site; Trust; United States; Viral; Virus
MeSH Terms: conditions — Hepatitis C; Medication Adherence; Behavior, Addictive; Hepatitis C, Chronic; Directly Observed Therapy; Disease; Infections; Liver Diseases; Liver Failure; Mental Disorders; Virus Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Modified Directly Observed Therapy (mDOT) (Experimental): In our mDOT model, pegylated interferon is administered once weekly, and one daily dose of oral medication is administered at the methadone window.
  Interventions: Other: Intensive Models (mDOT and CGT) of HCV Care
- Concurrent Group Treatment (CGT) (Experimental): In our CGT model, patients initiate HCV treatment within a once weekly treatment group which provides social support to mitigate fears of side effects, promote efficient education, and deliver weekly injections.
  Interventions: Other: Intensive Models (mDOT and CGT) of HCV Care
- Treatment as Usual (Active Comparator): In the TAU arm, subjects will receive all medications monthly (or more often as needed) at the clinic.
  Interventions: Other: Intensive Models (mDOT and CGT) of HCV Care

INTERVENTIONS:
Other: Intensive Models (mDOT and CGT) of HCV Care — Modified Directly Observed therapy (mDOT) and concurrent group treatment (CGT) are on-site HCV treatment models.

SUMMARY:
Injection drug users (IDUs) constitute 60% of the approximately 5 million people in the U.S. infected with hepatitis C virus (HCV). HCV treatment leading to sustained viral response (SVR) is associated with increased survival. However, IDUs have had poor access to HCV care and their success in HCV treatment has been limited. With direct-acting antiviral agents, HCV treatment delivered within large clinical trials leads to SVR or cure in over 70% of genotype-1 infected patients, compared to 45% with previous therapies. However, SVR rates are as low as 14% in real-world settings. The majority of patients who fail to achieve SVR will develop drug resistance, but the optimal adherence level to minimize resistance is unknown. If HCV treatment continues to be delivered within current models of care, most IDUs will not only fail treatment and develop resistance, but may transmit resistant viruses to others. We have previously developed a multidisciplinary model of HCV care which integrates on-site primary care, substance abuse treatment, psychiatric care, and HCV-related care within opiate agonist treatment clinics. To maximize treatment outcomes, we piloted two models of intensive HCV-related care: directly observed therapy (DOT), and concurrent group therapy (CGT). In our DOT model, pegylated interferon is administered once weekly, if applicable, and one daily dose of oral medication is administered at the methadone window. In our CGT model, patients initiate HCV treatment within a once weekly treatment group which provides powerful social support to mitigate fears of side effects, promote efficient education, and deliver weekly injections, if applicable. It is unknown whether either model is better or more cost-effective than standard on-site care.

PREVAIL 1: In the proposed study, 150 IDUs with chronic HCV (genotype 1) will be recruited from methadone clinics and randomized to one of three models of care: DOT; concurrent group treatment; or standard on-site care. Our specific aims are: 1) To determine whether either of two intensive on-site HCV treatment models (DOT or concurrent group treatment) is more efficacious than standard on-site treatment for enhancing adherence and SVR, and decreasing drug resistance; (2) To determine the incidence and factors associated with the development of drug resistance in IDUs; (3) To perform cost and cost-effectiveness analyses of each model; (4) To examine the impact of HIV coinfection on adherence and virologic outcomes among HCV-infected IDUs.

PREVAIL 2: In the proposed study, 60 IDUs with chronic HCV (genotypes 1 2, 3 and 4) will be recruited from opiate agonist treatment programs and started on HCV treatment. Subjects will be offered the choice of model of care (either standard on-site, DOT, or concurrent group treatment). Our specific aims are: (1) to determine rates of adherence and SVR in a cohort of opiate agonist treatment patients initiating treatment with sofosbuvir-based regimens and (2) to determine adherence rates over time in drug users (genotype 3 and genotype 1 / IFN-ineligible) initiating a 24 week IFN-free regimen.

PREVAIL 3: In the proposed study, 60 IDUs with chronic HCV (genotype 1 and 4) will be recruited from opiate agonist treatment programs and started on HCV treatment. Subjects will be offered the choice of model of care (either standard on-site, DOT, or concurrent group treatment). Our specific aims are: (1) to determine rates of adherence and SVR in a cohort of opiate agonist treatment patients initiating treatment with oral DAA combination of sofosbuvir and simeprevir or fixed dose of sofosbuvir and ledipasvir and (2) to determine adherence rates over time in drug users.

DETAILED DESCRIPTION:
PREVAIL 1: In the proposed study, 150 IDUs with chronic HCV (genotype 1) will be recruited from methadone clinics and randomized to one of three models of care: DOT; concurrent group treatment; or standard on-site care. Our specific aims are: 1) To determine whether either of two intensive on-site HCV treatment models (DOT or concurrent group treatment) is more efficacious than standard on-site treatment for enhancing adherence and SVR, and decreasing drug resistance; (2) To determine the incidence and factors associated with the development of drug resistance in IDUs; (3) To perform cost and cost-effectiveness analyses of each model; (4) To examine the impact of HIV coinfection on adherence and virologic outcomes among HCV-infected IDUs.

PREVAIL 2: In the proposed study, 60 IDUs with chronic HCV (genotypes 1 2, 3 and 4) will be recruited from opiate agonist treatment programs and started on HCV treatment. Subjects will be offered the choice of model of care (either standard on-site, DOT, or concurrent group treatment). Our specific aims are: (1) to determine rates of adherence and SVR in a cohort of opiate agonist treatment patients initiating treatment with sofosbuvir-based regimens and (2) to determine adherence rates over time in drug users (genotype 3 and genotype 1 / IFN-ineligible) initiating a 24 week IFN-free regimen.

PREVAIL 3: In the proposed study, 60 IDUs with chronic HCV (genotype 1 and 4) will be recruited from opiate agonist treatment programs and started on HCV treatment. Subjects will be offered the choice of model of care (either standard on-site, DOT, or concurrent group treatment). Our specific aims are: (1) to determine rates of adherence and SVR in a cohort of opiate agonist treatment patients initiating treatment with oral DAA combination of sofosbuvir and simeprevir or fixed dose of sofosbuvir and ledipasvir and (2) to determine adherence rates over time in drug users.

ELIGIBILITY:
Eligibility Ages Eligible for Study: 18 Years and older Genders Eligible for Study: Both

PREVAIL 1:

Inclusion Criteria:

* HCV-infected, Genotype-1
* Treatment naïve or treatment experienced patients
* Willing to receive HCV treatment on-site
* Initiating treatment with direct-acting antiviral agents (DAA) with or without ribavirin +/- pegylated interferon alfa-2a
* Receiving methadone or buprenorphine in clinic at least one time per week
* Age 18 or older
* Able to provide informed consent
* Psychiatrically stable
* English or Spanish speaking
* Currently enrolled in a methadone or buprenorphine treatment program in the designated clinics in the Bronx (Melrose, Port Morris, Waters Place)

Exclusion Criteria:

* Known hypersensitivity (allergy) to interferon, ribavirin or DAA
* Psychiatrically unstable
* Pregnant or breast-feeding

PREVAIL 2:

Inclusion Criteria:

* HCV-infected, Genotype-1, , 2, 3, or 4
* Willing to receive HCV treatment on-site at an opiate agonist treatment program.
* Initiating treatment with sofosbuvir and ribavirin +/- pegylated interferon alfa-2a
* Age 18 or older
* Able to provide informed consent
* English or Spanish speaking
* Currently a patient in one of the designated clinics in the Bronx (Melrose, Port Morris, Waters Place)

Exclusion Criteria:

* Known hypersensitivity (allergy) to interferon, ribavirin or sofosbuvir
* Pregnant or breast-feeding

PREVAIL 3:

Inclusion Criteria:

* HCV-infected, Genotype-1 or 4
* Willing to receive HCV treatment on-site at an opiate agonist treatment program.
* Initiating treatment with oral DAA combination of sofosbuvir and simeprevir or fixed dose of sofosbuvir and ledipasvir.
* Age 18 or older
* Able to provide informed consent
* English or Spanish speaking
* Currently a patient in one of the designated clinics in the Bronx (Melrose, Port Morris, Waters Place)

Exclusion Criteria:

* Known hypersensitivity (allergy) to sofosbuvir, simprevir or ledipasvir.
* Pregnant or breast-feeding

PREVAIL 4

Inclusion Criteria:

* HCV-infected, Genotype-1
* Treatment naïve or treatment experienced patients
* Willing to receive HCV treatment on-site
* Initiating treatment with direct-acting antiviral agents (DAA) with or without ribavirin +/- pegylated interferon alfa-2a
* Age 18 or older
* Able to provide informed consent
* Psychiatrically stable
* English or Spanish speaking

Exclusion Criteria:

* Known hypersensitivity (allergy) to interferon, ribavirin or DAA
* Psychiatrically unstable
* Pregnant or breast-feeding

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Actual)
Dates: Start 2013-10-01 (Actual); Primary Completion 2017-04-30 (Actual); Study Completion 2017-04-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Garland Gudger, MD, MPH, Principal Investigator — Prisma Health-Upstate
Locations (1):
- Greenville Health System, Greenville, South Carolina, United States

REFERENCES:
- [Derived] Heo M, Pericot-Valverde I, Rennert L, Akiyama MJ, Norton BL, Gormley M, Agyemang L, Arnsten JH, Litwin AH. Hepatitis C Virus Direct-Acting Antiviral Treatment Adherence Patterns and Sustained Viral Response Among People Who Inject Drugs Treated in Opioid Agonist Therapy Programs. Clin Infect Dis. 2021 Dec 6;73(11):2093-2100. doi: 10.1093/cid/ciab334. PMID 33876230
- [Derived] Pericot-Valverde I, Heo M, Akiyama MJ, Norton BL, Agyemang L, Niu J, Litwin AH. Factors and HCV treatment outcomes associated with smoking among people who inject drugs on opioid agonist treatment: secondary analysis of the PREVAIL randomized clinical trial. BMC Infect Dis. 2020 Dec 4;20(1):928. doi: 10.1186/s12879-020-05667-3. PMID 33276738
- [Derived] Akiyama MJ, Norton BL, Arnsten JH, Agyemang L, Heo M, Litwin AH. Intensive Models of Hepatitis C Care for People Who Inject Drugs Receiving Opioid Agonist Therapy: A Randomized Controlled Trial. Ann Intern Med. 2019 May 7;170(9):594-603. doi: 10.7326/M18-1715. Epub 2019 Apr 9. PMID 30959528
- [Derived] Akiyama MJ, Agyemang L, Arnsten JH, Heo M, Norton BL, Schackman BR, Linas BP, Litwin AH. Rationale, design, and methodology of a trial evaluating three models of care for HCV treatment among injection drug users on opioid agonist therapy. BMC Infect Dis. 2018 Feb 9;18(1):74. doi: 10.1186/s12879-018-2964-5. PMID 29426304

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Hepatitis C virus-infected PWID from 3 OAT programs in Bronx, New York, were enrolled beginning in October 2013, and participants were followed until April 2017. Potential participants were referred by clinicians if they were eligible for HCV treatment on the basis of guidelines from the American Association for the Study of Liver Diseases and Infectious Diseases Society of America (AASLD/IDSA). Eligibility was assessed by an oral screener and a confirmatory chart review.
Period: Overall Study
Arm/Group | Modified Directly Observed Therapy (mDOT) | Concurrent Group Treatment (CGT) | Treatment as Usual
Started | 51 | 48 | 51
Completed | 51 | 48 | 51 (Three SIT participants with no available blister pack adherence data were not included in the analysis of the primary adherence outcome.)
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Modified Directly Observed Therapy (mDOT) | Concurrent Group Treatment (CGT) | Treatment as Usual | Total
Number analyzed (Participants) | 51 | 48 | 51 | 150
Age, Continuous [Mean (Standard Deviation); unit: Years] | 51.4 (10) | 51.2 (11) | 51.0 (11) | 51.2 (11)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 18 | 16 | 19 | 53
  Male | 33 | 32 | 32 | 97
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 31 | 24 | 29 | 84
  Not Hispanic or Latino | 20 | 24 | 22 | 66
  Unknown or Not Reported | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 3 | 1 | 5
  Asian | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 1 | 1
  Black or African American | 12 | 13 | 13 | 38
  White | 6 | 5 | 4 | 15
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 32 | 27 | 32 | 91
Region of Enrollment [Number; unit: participants]
  United States | 51 | 48 | 51 | 150
Homelessness [Count of Participants; unit: Participants]
  Homeless | 9 | 10 | 15 | 34
  Housed | 42 | 38 | 36 | 116
Employment Status [Count of Participants; unit: Participants]
  Employed | 8 | 10 | 10 | 28
  Unemployed | 43 | 38 | 41 | 122
Marital Status [Count of Participants; unit: Participants]
  Married (Living with partner) | 18 | 21 | 16 | 55
  Not Married | 33 | 27 | 35 | 95
Urine Drug Screen (6 mo before baseline) [Number; unit: Number of participants] — Urine drug screen results for participants within 6 months of baseline visit. Participant count indicates those who tested positive for the indicated substance.
  Number of participants
    Any Drug | 34 | 34 | 30 | 98
    Opioids | 23 | 26 | 21 | 70
    Cocaine | 24 | 23 | 24 | 71
    Benzodiazepines | 15 | 15 | 13 | 43
Self-Reported Durg Use (30 days before baseline) [Number; unit: Participants] — Measure Description: Urine drug screen results for participants within 30 days of baseline visit. Participant count indicates those who tested positive for the indicated substance.
  Participants
    Heroin | 9 | 9 | 10 | 28
    Other opioids/analgesics | 10 | 8 | 15 | 33
    Cocaine | 12 | 12 | 12 | 36
    Sedative/hypnotics/tranquilizers | 9 | 12 | 12 | 33
    Amphetamines | 3 | 0 | 1 | 4
Alcohol use to intoxication (30 days before baseline) [Count of Participants; unit: Participants] | 13 | 11 | 12 | 36
Injection drug use [Count of Participants; unit: Participants] | 38 | 40 | 35 | 113
Comorbid psychiatric conditions [Number; unit: participants]
  Any | 20 | 22 | 25 | 67
  Major depressive episode | 11 | 15 | 12 | 38
  Generalized anxiety disorder | 8 | 10 | 10 | 28
  Psychotic disorder | 12 | 17 | 20 | 49
  Current manic episode | 1 | 6 | 4 | 11
Depression (PHQ-9) [Count of Participants; unit: Participants]
  None or mild | 33 | 33 | 31 | 97
  Moderate or severe | 18 | 15 | 20 | 53
HIV/HCV co-infection [Count of Participants; unit: Participants] | 6 | 6 | 9 | 21
HCV subtype [Number; unit: participants] — Subtype determined by medical chart review
  participants
    1a | 43 | 41 | 44 | 128
    1b | 8 | 7 | 7 | 22
Cirrhosis [Count of Participants; unit: Participants] | 15 | 16 | 10 | 41
Treatment experienced [Count of Participants; unit: Participants] | 43 | 6 | 6 | 55
DAA regimen [Count of Participants; unit: Participants] — Direct acting antivirals (DAA) are medication for treating HCV. Several drug combinations were used to treat participants in this study and are listed here.
  Participants
    SOF/LDV | 31 | 38 | 35 | 104
    SOF/SMV | 5 | 2 | 4 | 11
    SOF/RBV | 9 | 3 | 5 | 17
    SOF/IFN/RBV | 5 | 3 | 7 | 15
    TVR/IFN/RBV | 1 | 2 | 0 | 3
Opioid agonist therapy [Number; unit: participants]
  Methadone | 51 | 47 | 49 | 147
  Buprenorphine | 0 | 1 | 2 | 3
Opioid agonist pick-up schedule [Count of Participants; unit: Participants]
  1-3 per week | 6 | 12 | 14 | 32
  4-6 per week | 45 | 36 | 37 | 118
Urine drug screen (at baseline) [Number; unit: participants] — Measure Description: Urine drug screen results for participants at baseline visit. Participant count indicates those who tested positive for the indicated substance.
  participants
    Any drug | 26 | 23 | 25 | 74
    Opioids/oxycodone | 12 | 14 | 11 | 37
    Cocaine | 17 | 11 | 16 | 44
    Benzodiazepines | 9 | 4 | 10 | 23
    Amphetamines | 0 | 0 | 0 | 0
IL28B Genotype [Count of Participants; unit: Participants] — Genotype was determined through medical record chart review.
  Participants
    CC | 9 | 11 | 13 | 33
    TC | 26 | 26 | 27 | 79
    TT | 16 | 11 | 11 | 38

OUTCOME MEASURES:

1. Primary Outcome: Electronically Monitored Medication Adherence
Description: Hepatitis C medication adherence will be measured using electronic blister pack monitoring.
Time Frame: 1-12 weeks
Measure: Mean (95% Confidence Interval); unit: Percentage of medication taken
Arm/Group | Modified Directly Observed Therapy (mDOT) | Concurrent Group Treatment (CGT) | Treatment as Usual
Number analyzed (Participants) | 51 | 48 | 51
Percentage of medication taken | 86 [80 to 92] | 80 [74 to 86] | 75 [70 to 81]

2. Secondary Outcome: Sustained Virologic Response
Description: Undetectable HCV RNA at posttreatment week 12.
Time Frame: 12 weeks after treatment completion
Measure: Count of Participants; unit: Participants
Arm/Group | Modified Directly Observed Therapy (mDOT) | Concurrent Group Treatment (CGT) | Treatment as Usual
Number analyzed (Participants) | 51 | 48 | 51
Participants | 50 | 45 | 46

3. Secondary Outcome: HCV Treatment Completion
Description: Completion of ≥80% of the planned treatment course. For example, ≥10 wk of a 12-wk course, or ≥20 wk of a 24-wk course.
Time Frame: Up to 48 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Modified Directly Observed Therapy (mDOT) | Concurrent Group Treatment (CGT) | Treatment as Usual
Number analyzed (Participants) | 51 | 48 | 51
Participants | 50 | 47 | 48

ADVERSE EVENTS:
Time Frame: 8 months / 36 weeks
Arm/Group | Modified Directly Observed Therapy (mDOT) | Concurrent Group Treatment (CGT) | Treatment as Usual
All-Cause Mortality (participants affected / at risk) | 0/51 | 1/48 | 1/51
Serious Adverse Events (participants affected / at risk) | 0/51 | 0/48 | 0/51
Other Adverse Events (participants affected / at risk) | 1/51 | 3/48 | 5/51
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Modified Directly Observed Therapy (mDOT) (N=51) | Concurrent Group Treatment (CGT) (N=48) | Treatment as Usual (N=51)
Virologic Failure (HCV) (Hepatobiliary disorders) | 1 (1) | 3 (3) | 5 (5)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2012-09-01): https://cdn.clinicaltrials.gov/large-docs/45/NCT01857245/Prot_SAP_000.pdf